CLINICAL TRIAL: NCT03053453
Title: Evaluation of the Patient Reported Outcomes After Sensor-guided Total Knee Arthroplasty Under Spinal Anesthesia With Limited Motor-block.
Brief Title: Evaluation of Patient Reported Outcomes (PRO) After Total Knee Arthroplasty (TKA) Under Spinal Anesthesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of study surgeon investigator.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00129
Record Dates: First submitted 2017-01-30; First posted 2017-02-15 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Knee Injuries
Keywords: Total Knee Replacement Arthroplasty
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomized prospective study looking at the impact sensor guidance has on the outcome of patients and comparing to that of patients with a standard technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Spinal Surgery (Active Comparator): Patients will be given spinal anesthesia with 2.6 mL of 0.5% isobaric bupivacaine.
  Interventions: Procedure: Spinal Surgery
- Sensor Guided Spinal Surgery (Experimental): The Verasense Knee System device (OrthoSensor inc., Dania Beach, Florida) is a sterile sensor system that replaces the tibial insert trials used during surgery. The sensor contains a microprocessor and integrated nanosensor system, which wirelessly transmits real-time data to a portable graphic display unit used for read-out of the data. The sensor measures and localizes peak load at the medial and lateral tibiofemoral joint interfaces. Loading data is thereby captured intra-operatively through the full range of movement (ROM) using the sensor system.
  Interventions: Device: Verasense Knee System device

INTERVENTIONS:
Procedure: Spinal Surgery — TKA under standard of care spinal surgery.
  Arms: Standard of Care Spinal Surgery
Device: Verasense Knee System device — Sensor measures and localizes peak load at the medial and lateral tibiofemoral joint interfaces. Loading data is thereby captured intra-operatively through the full range of movement (ROM) using the sensor system.
  Other Names: OrthoSensor
  Arms: Sensor Guided Spinal Surgery

SUMMARY:
The purpose of this study will be to evaluate and compare patients undergoing total knee arthroplasty (TKA) with sensor guidance versus that of a standard technique. Each patient will be assessed for the difference between passive, soft tissue controlled, pressure balance and muscle activated pressure balance.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be screened for eligibility based on whether they have chronic knee pain as a result of an arthritis-related condition.
* Patient with chronic knee pain who is indicated for total hip or knee replacement surgery
* Patient is at least 50 years of age
* Patient is willing to participate in pre- and postoperative surveys

Exclusion Criteria:

* Failure to complete pre-operative surveys.
* Revision Total Knee Arthroplasty
* Prior ipsilateral knee surgery such as ligament reconstruction or osteotomy
* Contralateral Total Knee Arthroplasty
* Prior tibial plateau fracture
* Ligamentous Insufficiency
* History of fibromyalgia, chronic fatigue syndrome

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hertling, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Spinal Surgery | Sensor Guided Spinal Surgery
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study personnel involved in data collection did not log information on patients in the Standard of Care Spinal Surgery Arm into the study's shared drive. These personnel have since departed from the institution. All efforts by the study team to obtain this information/contact the departed personnel have been unsuccessful. The Principal Investigator believes these missing data to be permanently unavailable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Spinal Surgery | Sensor Guided Spinal Surgery | Total
Number analyzed (Participants) | 0 | 26 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 71.3 (7.1) | 71.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 15 | 15
  Male |  | 11 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 18 | 18
  Unknown or Not Reported |  | 8 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 24 | 24
  More than one race |  | 1 | 1
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 26 | 26

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score (KSS)
Description: The Knee Society Score (KSS) comprises two sections (each worth 100 points) for a maximum 200 points. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. For each section, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.
Time Frame: Month 12 Post-Surgery
Population: This study was interrupted as the surgeon investigator decided to retire from clinical practice. Following the surgeon investigator's assessment, no intervention was performed based on the intra-operative results of the pressure load measurement. For that reason, the PI deemed the study team should not compare the surgical results using the KSS. Therefore, this measure was not assessed among study participants; no data are available for this outcome measure as it was not assessed.
Arm/Group | Standard of Care Spinal Surgery | Sensor Guided Spinal Surgery
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, function in daily living (ADLs), sports/recreation, and quality of life. The maximum score a patient can achieve is 100, indicating no knee problems. The minimum score is zero, indicating severe knee problems.
Time Frame: Month 12 Post-Surgery
Population: This study was interrupted as the surgeon investigator decided to retire from clinical practice. Following the surgeon investigator's assessment, no intervention was performed based on the intra-operative results of the pressure load measurement. For that reason, the PI deemed the study team should not compare the surgical results using the KOOS. Therefore, this measure was not assessed among study participants; no data are available for this outcome measure as it was not assessed.
Arm/Group | Standard of Care Spinal Surgery | Sensor Guided Spinal Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Description: Assessments performed by study personnel and surgical team while in the hospital; then assessments performed by surgeon at scheduled follow-up visits
Arm/Group | Standard of Care Spinal Surgery | Sensor Guided Spinal Surgery
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT03053453/Prot_000.pdf